CLINICAL TRIAL: NCT04056871
Title: Comparing the Association of Different Frailty Scores to the Incidence of Post-operative Delirium and Cognitive Dysfunction
Brief Title: Different Frailty Scores to Incidence of Post-operative Delirium and Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Loh Pui San, Consultant Anaesthesiologist, University of Malaya
Other Study IDs: U1111-1237-9788
Record Dates: First submitted 2019-08-08; First posted 2019-08-14 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Frail Elderly Syndrome; Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: post-operative delirium; post-operative cognitive dysfunction; frailty; nutritional status; depression
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Frailty; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fried Frailty Phenotype: This group of patients will be assess by using 5 characteristics of Frailty which are weight loss, weakness, exhaustion, low activity and physical fitness of the patients. Patients classify as frail will have more than 3 criteria, intermediate or pre-frail will be 1 or 2 criteria present and robust will not have criteria.
  Interventions: Diagnostic Test: Frailty Screening Tools
- Groningen Frailty Index: GFI is a simple questionnaire consisting of 15 items which are classified into 8 groups, consistent of 4 domains of functioning. A score of 4 or more indicates a higher risk for frailty and possible delirium.
  Interventions: Diagnostic Test: Frailty Screening Tools

INTERVENTIONS:
Diagnostic Test: Frailty Screening Tools — This is an observational and prospective study of patients who are going for elective surgery, thus no intervention will be given.

SUMMARY:
Patients who are frail will have higher rate for post-operative morbidities, mortality, prolonged hospital stays, loss of independence, increase in institutionalization, post-operative cognitive dysfunction (POCD) and delirium (POD).

So, it is crucial to find a suitable frailty assessment tool that can be incorporated into a guideline and reference for our local setting in geriatric peri-operative management. In the mean time, create awareness regarding the frailty elderly population with POD, POCD and other associated poor outcomes among our clinicians.

DETAILED DESCRIPTION:
Increasing life expectancy has led to increase in elderly populations, thus the elderly patients amounting for greater proportion of surgical cases. But, most of them are frail with multiple co-morbidities and are exposed to adverse outcome post-operatively. The commonest adverse outcomes is post-operative delirium (POD) in which clinicians often miss and often take lightly. If it is not treated, it will progress to post-operative cognitive dysfunction (POCD).

So, it is crucial to identify the risk factors pre-operatively to minimize the risk of POD and POCD. The frail patients are more likely to have pre-existing cognitive impairment with reduced cognitive reserve, hence, they are the most vulnerable to POCD and POD. One of the most commonly used frailty screening tools is Fried Frailty criteria which is an easily accessible tool that mainly screens and scores the patients physically. However, the investigators propose to use the Groningen Frailty scale as it can assess the patients in a more holistic approach, not only in physical, but also vision, heating, nutritional, co-morbidities, cognition, psychosocial and mobility of the patients.

Method:

Elderly patients >65 years old undergoing elective surgery under general or local anaesthesia in University Malaya Medical Centre will be recruited for this study, over a 6 months period from August 2019 to January 2020. Patients will be assessed with baseline cognitive assessment, nutritional status, psychological status, and frailty scores prior to the surgery. After the operation, patients will be assessed using 4AT and CAM for at least 5 days or until patients discharged. Cognitive functions will be assessed on post-operative 7th day, 1 month and 3 months with T-MOCA via phone.

All data will be analyzed using SPSS.

Impact of research:

A suitable frailty assessment tool will be identified to be used pre-operatively for elderly patients undergoing elective surgery. This tool will then be incorporated into a guideline and reference in our local setting for geriatric peri-operative management protocol.

Moreover, with the results, investigators hope to create awareness within our multidisciplinary care of elderly surgical population on frailty assessment and its correlation to post-operative delirium, cognitive dysfunction and associated poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years old and above
* ASA 1 - 3
* Full GCS
* Elective surgery
* Able to communicate well
* Consented
* Extubated at the end of surgery

Exclusion Criteria:

* Cardiac and neurosurgery
* On drugs affecting the central nervous system
* Admission to ICU intubated to continue ventilation.
* Refusal of consent
* Severe hearing loss
* Unable to use telephone/ mobile phone for communication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients above 65 years of age undergoing elective surgery under anesthetic care for both general and regional anesthesia with or without sedation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Occurence of confusion using Confusion Assessment Method (CAM) scores | Within 5 days after surgery
  Delirium is present if the following are present:
  Feature 1-Acute Change or/and Fluctuation (any symptom) AND Feature 2-Inattention AND EITHER Feature 3-Disorganized Thinking OR Feature 4-Altered Level of Consciousness
Change in cognitive function using Telephone-Montreal Cognitive Assessment (T-MOCA) | Within 1 month
  Cognitive function of the patients will be assessed after discharged and must achieved post-operative day 7 with T-MOCA via phone, subsequently assessed at 1 month and 3 month later.
Occurence of delirium using 4AT scores | Within 5 days after surgery
  A score of 4 or more suggests delirium but is not diagnostic: more detailed assessment of mental status may be required to reach a diagnosis. A score of 1-3 suggests cognitive impairment and more detailed cognitive testing and informant history-taking are required. A score of 0 does not definitively exclude delirium or cognitive impairment: more detailed testing may be required depending on the clinical context.

CONTACTS AND LOCATIONS:
Overall Officials: Pui San Loh, Principal Investigator — University of Malaya
Locations (1):
- University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718
- [Background] Peri-operative Care for Older Patients Undergoing Surgery. British Geriatrics Society. http://www.bgs.org.uk/index.php/topresources/publicationfind/goodpractice/2402-bpg-pops (cited November 2015
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Collard RM, Boter H, Schoevers RA, Oude Voshaar RC. Prevalence of frailty in community-dwelling older persons: a systematic review. J Am Geriatr Soc. 2012 Aug;60(8):1487-92. doi: 10.1111/j.1532-5415.2012.04054.x. Epub 2012 Aug 6. PMID 22881367
- [Background] Fried LP, Xue QL, Cappola AR, Ferrucci L, Chaves P, Varadhan R, Guralnik JM, Leng SX, Semba RD, Walston JD, Blaum CS, Bandeen-Roche K. Nonlinear multisystem physiological dysregulation associated with frailty in older women: implications for etiology and treatment. J Gerontol A Biol Sci Med Sci. 2009 Oct;64(10):1049-57. doi: 10.1093/gerona/glp076. Epub 2009 Jun 30. PMID 19567825
- [Background] Sepehri A, Beggs T, Hassan A, Rigatto C, Shaw-Daigle C, Tangri N, Arora RC. The impact of frailty on outcomes after cardiac surgery: a systematic review. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3110-7. doi: 10.1016/j.jtcvs.2014.07.087. Epub 2014 Aug 7. PMID 25199821
- [Background] Beggs T, Sepehri A, Szwajcer A, Tangri N, Arora RC. Frailty and perioperative outcomes: a narrative review. Can J Anaesth. 2015 Feb;62(2):143-57. doi: 10.1007/s12630-014-0273-z. Epub 2014 Nov 25. PMID 25420470
- [Background] Desserud KF, Veen T, Soreide K. Emergency general surgery in the geriatric patient. Br J Surg. 2016 Jan;103(2):e52-61. doi: 10.1002/bjs.10044. Epub 2015 Dec 1. PMID 26620724
- [Background] Lin HS, McBride RL, Hubbard RE. Frailty and anesthesia - risks during and post-surgery. Local Reg Anesth. 2018 Oct 5;11:61-73. doi: 10.2147/LRA.S142996. eCollection 2018. PMID 30323657
- [Background] Dasgupta M, Dumbrell AC. Preoperative risk assessment for delirium after noncardiac surgery: a systematic review. J Am Geriatr Soc. 2006 Oct;54(10):1578-89. doi: 10.1111/j.1532-5415.2006.00893.x. PMID 17038078
- [Background] Peters LL, Boter H, Buskens E, Slaets JP. Measurement properties of the Groningen Frailty Indicator in home-dwelling and institutionalized elderly people. J Am Med Dir Assoc. 2012 Jul;13(6):546-51. doi: 10.1016/j.jamda.2012.04.007. Epub 2012 May 12. PMID 22579590
- [Background] Bielderman A, van der Schans CP, van Lieshout MR, de Greef MH, Boersma F, Krijnen WP, Steverink N. Multidimensional structure of the Groningen Frailty Indicator in community-dwelling older people. BMC Geriatr. 2013 Aug 22;13:86. doi: 10.1186/1471-2318-13-86. PMID 23968433
- [Background] Steverink N, Slaets J, Schuurmans H, van Lis M. Measuring frailty: developing and testing of the Groningen frailty indicator (GFI). Gerontologist. 2001;41:236-237
- [Background] Shem Tov L, Matot I. Frailty and anesthesia. Curr Opin Anaesthesiol. 2017 Jun;30(3):409-417. doi: 10.1097/ACO.0000000000000456. PMID 28291129
- [Background] Lin HS, Watts JN, Peel NM, Hubbard RE. Frailty and post-operative outcomes in older surgical patients: a systematic review. BMC Geriatr. 2016 Aug 31;16(1):157. doi: 10.1186/s12877-016-0329-8. PMID 27580947
- [Background] Oakland K, Nadler R, Cresswell L, Jackson D, Coughlin PA. Systematic review and meta-analysis of the association between frailty and outcome in surgical patients. Ann R Coll Surg Engl. 2016 Feb;98(2):80-5. doi: 10.1308/rcsann.2016.0048. Epub 2016 Jan 7. PMID 26741674
- [Background] Buigues C, Juarros-Folgado P, Fernandez-Garrido J, Navarro-Martinez R, Cauli O. Frailty syndrome and pre-operative risk evaluation: A systematic review. Arch Gerontol Geriatr. 2015 Nov-Dec;61(3):309-21. doi: 10.1016/j.archger.2015.08.002. Epub 2015 Aug 4. PMID 26272286
- [Background] Hogue CW Jr, Palin CA, Arrowsmith JE. Cardiopulmonary bypass management and neurologic outcomes: an evidence-based appraisal of current practices. Anesth Analg. 2006 Jul;103(1):21-37. doi: 10.1213/01.ANE.0000220035.82989.79. PMID 16790619
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Pendlebury ST, Welch SJ, Cuthbertson FC, Mariz J, Mehta Z, Rothwell PM. Telephone assessment of cognition after transient ischemic attack and stroke: modified telephone interview of cognitive status and telephone Montreal Cognitive Assessment versus face-to-face Montreal Cognitive Assessment and neuropsychological battery. Stroke. 2013 Jan;44(1):227-9. doi: 10.1161/STROKEAHA.112.673384. Epub 2012 Nov 8. PMID 23138443
- [Background] Ismail Z, Rajji TK, Shulman KI. Brief cognitive screening instruments: an update. Int J Geriatr Psychiatry. 2010 Feb;25(2):111-20. doi: 10.1002/gps.2306. PMID 19582756
- [Background] Robinson TN, Wu DS, Pointer LF, Dunn CL, Moss M. Preoperative cognitive dysfunction is related to adverse postoperative outcomes in the elderly. J Am Coll Surg. 2012 Jul;215(1):12-7; discussion 17-8. doi: 10.1016/j.jamcollsurg.2012.02.007. Epub 2012 May 22. PMID 22626912
- [Background] Polanczyk CA, Marcantonio E, Goldman L, Rohde LE, Orav J, Mangione CM, Lee TH. Impact of age on perioperative complications and length of stay in patients undergoing noncardiac surgery. Ann Intern Med. 2001 Apr 17;134(8):637-43. doi: 10.7326/0003-4819-134-8-200104170-00008. PMID 11304103
- [Background] Hamel MB, Henderson WG, Khuri SF, Daley J. Surgical outcomes for patients aged 80 and older: morbidity and mortality from major noncardiac surgery. J Am Geriatr Soc. 2005 Mar;53(3):424-9. doi: 10.1111/j.1532-5415.2005.53159.x. PMID 15743284
- [Background] Etzioni DA, Liu JH, O'Connell JB, Maggard MA, Ko CY. Elderly patients in surgical workloads: a population-based analysis. Am Surg. 2003 Nov;69(11):961-5. PMID 14627256
- [Background] Moug SJ, Stechman M, McCarthy K, Pearce L, Myint PK, Hewitt J; Older Persons Surgical Outcomes Collaboration. Frailty and cognitive impairment: Unique challenges in the older emergency surgical patient. Ann R Coll Surg Engl. 2016 Mar;98(3):165-9. doi: 10.1308/rcsann.2016.0087. PMID 26890834
- [Background] Verloo H, Goulet C, Morin D, von Gunten A. Association between frailty and delirium in older adult patients discharged from hospital. Clin Interv Aging. 2016 Jan 18;11:55-63. doi: 10.2147/CIA.S100576. eCollection 2016. PMID 26848261
- [Background] Hamilton GM, Wheeler K, Di Michele J, Lalu MM, McIsaac DI. A Systematic Review and Meta-analysis Examining the Impact of Incident Postoperative Delirium on Mortality. Anesthesiology. 2017 Jul;127(1):78-88. doi: 10.1097/ALN.0000000000001660. PMID 28459734
- [Background] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844
- [Background] Inouye SK, Charpentier PA. Precipitating factors for delirium in hospitalized elderly persons. Predictive model and interrelationship with baseline vulnerability. JAMA. 1996 Mar 20;275(11):852-7. PMID 8596223
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Heymann A, Radtke F, Schiemann A, Lutz A, MacGuill M, Wernecke KD, Spies C. Delayed treatment of delirium increases mortality rate in intensive care unit patients. J Int Med Res. 2010 Sep-Oct;38(5):1584-95. doi: 10.1177/147323001003800503. PMID 21309472
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Radtke FM, Franck M, Schneider M, Luetz A, Seeling M, Heinz A, Wernecke KD, Spies CD. Comparison of three scores to screen for delirium in the recovery room. Br J Anaesth. 2008 Sep;101(3):338-43. doi: 10.1093/bja/aen193. Epub 2008 Jul 3. PMID 18603528
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Collins N, Blanchard MR, Tookman A, Sampson EL. Detection of delirium in the acute hospital. Age Ageing. 2010 Jan;39(1):131-5. doi: 10.1093/ageing/afp201. Epub 2009 Nov 16. No abstract available. PMID 19917632
- [Background] Kakuma R, du Fort GG, Arsenault L, Perrault A, Platt RW, Monette J, Moride Y, Wolfson C. Delirium in older emergency department patients discharged home: effect on survival. J Am Geriatr Soc. 2003 Apr;51(4):443-50. doi: 10.1046/j.1532-5415.2003.51151.x. PMID 12657062
- [Background] Bellelli G, Magnifico F, Trabucchi M. Outcomes at 12 months in a population of elderly patients discharged from a rehabilitation unit. J Am Med Dir Assoc. 2008 Jan;9(1):55-64. doi: 10.1016/j.jamda.2007.09.009. PMID 18187114
- [Background] Partridge JS, Martin FC, Harari D, Dhesi JK. The delirium experience: what is the effect on patients, relatives and staff and what can be done to modify this? Int J Geriatr Psychiatry. 2013 Aug;28(8):804-12. doi: 10.1002/gps.3900. Epub 2012 Oct 30. PMID 23112139
- [Background] Rockwood K. Educational interventions in delirium. Dement Geriatr Cogn Disord. 1999 Sep-Oct;10(5):426-9. doi: 10.1159/000017183. PMID 10473952
- [Background] Elie M, Rousseau F, Cole M, Primeau F, McCusker J, Bellavance F. Prevalence and detection of delirium in elderly emergency department patients. CMAJ. 2000 Oct 17;163(8):977-81. PMID 11068569
- [Background] Bellelli G, Morandi A, Davis DH, Mazzola P, Turco R, Gentile S, Ryan T, Cash H, Guerini F, Torpilliesi T, Del Santo F, Trabucchi M, Annoni G, Maclullich AM. Corrigendum to 'Validation of the 4AT, a new instrument for rapid delirium screening: a study in 234 hospitalised older people'. Age Ageing. 2015 Jan;44(1):175. doi: 10.1093/ageing/afu181. No abstract available. PMID 25477307
- [Background] de Vries NM, Staal JB, van Ravensberg CD, Hobbelen JS, Olde Rikkert MG, Nijhuis-van der Sanden MW. Outcome instruments to measure frailty: a systematic review. Ageing Res Rev. 2011 Jan;10(1):104-14. doi: 10.1016/j.arr.2010.09.001. Epub 2010 Sep 17. PMID 20850567
- [Background] Slaets JP. Vulnerability in the elderly: frailty. Med Clin North Am. 2006 Jul;90(4):593-601. doi: 10.1016/j.mcna.2006.05.008. PMID 16843764
- [Background] Fulop T, Larbi A, Witkowski JM, McElhaney J, Loeb M, Mitnitski A, Pawelec G. Aging, frailty and age-related diseases. Biogerontology. 2010 Oct;11(5):547-63. doi: 10.1007/s10522-010-9287-2. Epub 2010 Jun 18. PMID 20559726
- [Background] Walston J, Hadley EC, Ferrucci L, Guralnik JM, Newman AB, Studenski SA, Ershler WB, Harris T, Fried LP. Research agenda for frailty in older adults: toward a better understanding of physiology and etiology: summary from the American Geriatrics Society/National Institute on Aging Research Conference on Frailty in Older Adults. J Am Geriatr Soc. 2006 Jun;54(6):991-1001. doi: 10.1111/j.1532-5415.2006.00745.x. PMID 16776798
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Jones DM, Song X, Rockwood K. Operationalizing a frailty index from a standardized comprehensive geriatric assessment. J Am Geriatr Soc. 2004 Nov;52(11):1929-33. doi: 10.1111/j.1532-5415.2004.52521.x. PMID 15507074
- [Background] Mitnitski AB, Mogilner AJ, Rockwood K. Accumulation of deficits as a proxy measure of aging. ScientificWorldJournal. 2001 Aug 8;1:323-36. doi: 10.1100/tsw.2001.58. PMID 12806071
- [Background] Markle-Reid M, Browne G. Conceptualizations of frailty in relation to older adults. J Adv Nurs. 2003 Oct;44(1):58-68. doi: 10.1046/j.1365-2648.2003.02767.x. PMID 12956670
- [Background] Gobbens RJ, Luijkx KG, Wijnen-Sponselee MT, Schols JM. Toward a conceptual definition of frail community dwelling older people. Nurs Outlook. 2010 Mar-Apr;58(2):76-86. doi: 10.1016/j.outlook.2009.09.005. PMID 20362776